CLINICAL TRIAL: NCT03844932
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of ST-0529 in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study Evaluating the Efficacy and Safety of ST-0529 in Subjects With Moderately to Severely Active Ulcerative Colitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sublimity Board of Directors carefully evaluated the IA data: the 9.6% treatment remission difference for 75mg BID vs placebo (due to an increase in placebo response rate) was determined not sufficient to continue to fund the study
Sponsor: Sublimity Therapeutics Holdco Limited (Industry)
Collaborators: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CYC-202
Record Dates: First submitted 2019-01-31; First posted 2019-02-19 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: The study will investigate ST-0529 doses of 18.75 mg BID, 37.5 mg BID, or 75 mg BID, versus matching placebo BID.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be conducted as a double-blind study. Both the Investigator and subjects will be blinded with respect to the treatment the subject will receive. In addition, the central reader of the endoscopy assessment will be blinded to subject treatment for the entire study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ST-0529 18.75 mg* (Experimental): ST-0529: 18.75 mg orally twice daily (BID)
  *Jan 2021 update: following the IDMC recommendation, this arm has been dropped
  Interventions: Drug: ST-0529
- ST-0529 37.5 mg* (Experimental): ST-0529: 37.5 mg orally twice daily (BID)
  *Jan 2021 update: following the IDMC recommendation, this arm has been dropped
  Interventions: Drug: ST-0529
- ST-0529 75 mg (Experimental): ST-0529: 75 mg orally twice daily (BID)
  Interventions: Drug: ST-0529
- Matching Placebo (Placebo Comparator): Placebo: matching placebo orally twice daily (BID)
  Interventions: Drug: ST-0529

INTERVENTIONS:
Drug: ST-0529 — ST-0529 utilizes SmPill® technology to encapsulate the otherwise insoluble cyclosporine in a presolubilized, lipid-based formulation.
  Other Names: cyclosporine

SUMMARY:
Study CYC-202 is a multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of ST-0529 in subjects with moderately to severely active UC, defined as a score of 5 to 9 on the 3-Component Adapted Mayo Score (comprised of rectal bleeding, stool frequency and endoscopy sub-scores; score range 0-9).

DETAILED DESCRIPTION:
The study consists of a Screening period, Treatment period and Follow-up. The Screening period is comprised of two separate in-clinic visits, SV1 and SV2. At the initial Screening visit (SV1), subjects will be required to provide written informed consent to participate in the study and will then be assessed for eligibility. Electronic diaries will be provided to subjects at this visit to use for the duration of the study in order to record information relating to their UC disease. Subjects will return to the clinic for their Screening endoscopic assessment (SV2). Ulcerative colitis disease activity for eligibility will be assessed using the 3-Component Adapted Mayo Score. Upon successful completion of the Screening period, subjects will return to the clinic for their Baseline visit.

During the Treatment period, subjects will be evaluated in the clinic at Baseline (Day 1), Week 2, Week 4, Week 8, and Week 12 (End of Treatment Period). At Week 6 and Week 10, subjects will be contacted by telephone to assess Adverse Events (AEs), concomitant medication usage and study drug regimen adherence.

Subjects who complete the 12-week Treatment period will attend the Week 16 End of Study (EOS) visit. Subjects who discontinue study drug and withdraw or are withdrawn from the study before the Week 12 visit will be requested to return to the clinic as soon as possible to complete an Early Termination (ET) visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adult subjects 18 to 75 years old, inclusive.
2. Willing to provide written informed consent and to be compliant with the schedule of study visits and protocol assessments.
3. Diagnosis of UC established at least 3 months prior to the Baseline visit, by clinical and endoscopic evidence (colonoscopy or flexible sigmoidoscopy)
4. Moderately to severely active UC defined as the 3-Component Adapted Mayo Score of 5-9, inclusive, with an endoscopic sub-score of ≥ 2 (from central reading), and a rectal bleeding sub-score of ≥ 1, as determined 10 days (± 3 days) prior to Baseline.
5. Evidence of active UC, confirmed histologically (from local read), extending proximal to the rectum with ≥ 15 cm of involved colon.
6. At Screening, a colonoscopy will be required if the subject has had extensive colitis or pancolitis of > 8 years duration or left-sided colitis of > 12 years duration but has not had a colonoscopy within 1 year of the initial screening date. If the subject has had a colonoscopy within 1 year of the initial screening date, a flexible sigmoidoscopy may be used.
7. Subjects presenting at Screening with moderately to severely active UC demonstrating an inadequate response or loss of response or intolerance/medical contraindication to at least one of the following conventional therapies for UC:

   a. Corticosteroids:

   i. Signs and symptoms of active disease despite treatment with an adequate dose (e.g., prednisolone > 40 mg/day or equivalent) over a period of 4 weeks for oral therapy or intravenously (IV) for up to 1 week or ≥ 9 mg/day oral budesonide;

   OR

   ii. Unable to reduce corticosteroids below the equivalent of prednisolone 10 mg daily orally within 3 months of starting steroids or having experienced a relapse within 3 months of stopping steroids;

   OR

   iii. History of, or current intolerance to corticosteroids (including, but not limited to Cushing's syndrome, osteopenia/osteoporosis, hyperglycemia, insomnia, infection).

   b. Immunomodulators:

   i. Signs and symptoms of active disease despite at least 3 months of treatment with a sufficient dose (oral azathioprine ≥ 1.5 mg/kg or 6-mercaptopurine [6-MP] ≥ 0.75 mg/kg);

   OR

   ii. History of, or current dose-limiting toxicity associated with use of the agent (e.g., but not limited to nausea/vomiting, abdominal pain, pancreatitis, liver function test [LFT] abnormalities, lymphopenia, TPMT genetic mutation, infection).

   c. Anti-tumor necrosis factor (anti-TNF) agents:

   i. Signs and symptoms of active disease despite treatment with a single anti-TNF agent. Treatment failure is defined as a relapse after an initial response to therapy as follows:
   * Infliximab: At least 4 infusions of at least 5 mg/kg within a 14-week timeframe for induction and maintenance;
   * Adalimumab: Induction regimen incorporating 160 mg at Week 0 (four 40 mg injections in one day or two 40 mg injections per day for two consecutive days) and 80 mg at Week 2, followed by maintenance treatment of 40 mg every other week up to at least Week 8;
   * Golimumab: Induction regimen incorporating 200 mg subcutaneous (sc) injection at Week 0, followed by 100 mg at Week 2 and then maintenance treatment of 50 mg or 100 mg (weight dependent) every 4 weeks after completion of the induction regimen up to at least Week 12;

   OR

   ii. History of, or current intolerance (with an initial response), defined as the presence of clinically significant side-effects, including infusion-related hypersensitivity.

   d. Vedolizumab:

   i. Signs and symptoms of active disease despite a history of at least one induction regimen, defined as at least a 14-week (10 weeks in the EU) induction consisting of 300 mg IV at Weeks 0, 2 and 6.

   OR

   ii. History of intolerance to vedolizumab including, but not limited to, serious infections, hepatotoxicity, heart failure, allergic reactions, or any other condition that contributed to discontinuation of the agent.
8. Subjects receiving oral corticosteroids for the treatment of UC must be on a stable dose of ≤ 40 mg/day (prednisolone or equivalent), or ≤ 9 mg/day budesonide. This dose must be stable from the initial Screening visit until 1 week after the initiation of study treatment.
9. Subjects receiving oral 5-ASA must be on a stable dose from the initial Screening visit until the end of the study.
10. Subjects willing to cease the use of any therapeutic enema or suppository or foams, other than that required in preparation for study-mandated colonoscopy/flexible sigmoidoscopies, from the initial Screening visit until the end of the study.
11. Subjects willing to cease use of azathioprine or 6-MP from the initial Screening visit until the end of the study.
12. Negative serum pregnancy test in females of childbearing potential at Screening.
13. If female and of childbearing potential, must agree to be sexually abstinent or use one of the following highly effective methods of birth control from the initial Screening visit until 30 days after the last dose of study drug is administered:

    1. Hormonal contraceptives (e.g., combined oral contraceptives, patch, vaginal ring, injectables, and implants);
    2. Intrauterine contraceptive system;
    3. Surgical sterilization or partner sterile (must have documented proof);

    AND

    One of the following effective methods of birth control:
    1. Male/female condom;
    2. Cervical cap with spermicide;
    3. Diaphragm with spermicide;
    4. Contraceptive sponge.
14. Male subjects must be either surgically sterile (must have documented proof), agree to be sexually inactive or use a double-barrier method of birth control (e.g., condom and diaphragm with spermicide, condom with cervical cap and spermicide) from first study drug administration until 90 days after final drug administration.

Exclusion Criteria:

If a subject has any of the following criteria, they will be excluded from the study:

1. Subjects without previous treatment for UC.
2. Ulcerative colitis limited to rectum (ulcerative proctitis).
3. Evidence of acute severe colitis with toxic megacolon, abdominal abscess, bowel stricture or bowel perforation.
4. A diagnosis of Crohn's colitis, colitis yet to be classified, ischemic colitis, NSAID-induced colitis, idiopathic colitis (i.e., colitis not consistent with UC) or radiation colitis.
5. Subjects with evidence of pathogenic bowel infection (Clostridium difficile, Escherichia coli, Salmonella, Shigella or Campylobacter).
6. Previous surgery for UC or, in the opinion of the Investigator, will likely require surgery for UC during the study.
7. Any histological evidence of mucosal dysplasia.
8. Subjects with a current or recent history of severe, progressive or uncontrolled cardiac (including uncontrolled hypertension), renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurological (e.g., history of seizures) disease, abnormal magnesium or potassium levels, hypocholesterolemia, or any other severe co-morbidity that, in the opinion of the Investigator, could confound the study results or put the study subject at unreasonable risk.
9. Malignancies or history of malignancy within 5 years of the initial Screening visit, with the exception of adequately treated or excised non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin.
10. Any of the following laboratory abnormalities during the screening period - if values are initially outside the prescribed limits, the evaluation may be repeated once within the screening period to determine eligibility:

    1. Hemoglobin level < 8.0 g/dL
    2. Absolute WBC count < 3.0 × 10^9/L
    3. Absolute Lymphocyte count < 0.5 × 10^9/L
    4. Absolute neutrophil count < 1.2 × 10^9/L
    5. Platelet count < 100 × 10^9/L or >1200 × 10^9/L
    6. ALT or AST > 2.0 × ULN
    7. Alkaline phosphatase > 2.0 × ULN
    8. Serum creatinine > 1.5 × ULN
    9. Bilirubin > 1.5 × ULN
11. Subjects with active TB infection or known history of prior treated or untreated TB infection.
12. Subject with a positive serology test result for HIV (HIV type 1 or type 2).
13. Subject with a positive serology test result for active HBV or HCV infection.
14. Treatment with biologic agents for UC within 56 days or 5 half-lives (whichever is greater) prior to the Baseline visit.
15. Treatment with any calcineurin inhibitor (e.g. cyclosporine or tacrolimus) within 28 days prior to the Baseline visit.
16. Treatment with methotrexate or JAK inhibitors (e.g. tofacitinib) from the initial Screening visit until the end of the study.
17. Initiation of treatment with an oral or IV corticosteroid from the initial Screening visit until the end of the study.
18. Use of any strong inhibitors of CYP enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem, grapefruit juice and HIV antivirals) within 14 days prior to the Baseline visit.
19. Use of strong or moderate P-gp inhibitors (e.g., amiodarone, azithromycin, clarithromycin, itraconazole, ketoconazole, dronedarone, lapatinib, quinidine, ranolazine, verapamil) within 14 days prior to the Baseline visit.
20. Use of any herbal medication for the treatment of UC or which might interfere with CYP enzymes within 14 days prior to the Baseline visit.
21. Subjects vaccinated with a live or live-attenuated vaccine within 14 days of the Baseline visit, or planned vaccination during conduct of the study.
22. Subjects with a QTcF of > 450 ms for males and > 470 ms for females at Screening.
23. A history of risk factors for Torsades de pointes (e.g., history of heart failure, hypokalemia, family history of Long QT Syndrome).
24. Known hypersensitivity to cyclosporine or any excipients contained in ST-0529.
25. History of alcohol or drug abuse in the year prior to the initial Screening visit.
26. Subjects currently breast feeding, pregnant, or unwilling to delay initiation of breast feeding for at least 90 days after the last dose of study drug is administered.
27. Participation in another clinical trial and having received investigational medication within 30 days or within 5 half-lives (whichever is longer) prior to the Baseline visit, or concurrent participation in another clinical trial.
28. Subjects who, in the opinion of the Investigator, are unsuitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Clinical Remission at Week 12 | Week 12
  Stool frequency sub-score of ≤ 1 associated with a decrease ≥ 1 point from baseline, rectal bleeding sub-score of 0, and an endoscopic sub-score of ≤ 1 using the 3-Component Adapted Mayo Score.
  The 3-Component Adapted Mayo Score is a measure of UC disease ranging from 0 to 9 points and consists of 3 sub-scores, each graded from 0 - 3 with higher scores indicating more severe disease. The sub-scores are stool frequency (0 - 3); rectal bleeding (0 - 3); findings of endoscopy (0 - 3).

SECONDARY OUTCOMES:
Clinical Response at Week 12 | Week 12
  A decrease from baseline in the 3-Component Adapted Mayo Score of ≥ 2 points and ≥ 30%, with an accompanying decrease in the sub-score for rectal bleeding of ≥ 1 point or an absolute sub-score for rectal bleeding of ≤ 1.
  The 3-Component Adapted Mayo Score is a measure of UC disease ranging from 0 to 9 points and consists of 3 sub-scores, each graded from 0 - 3 with higher scores indicating more severe disease. The sub-scores are stool frequency (0 - 3); rectal bleeding (0 - 3); findings of endoscopy (0 - 3).
Endoscopic Healing at Week 12 | Week 12
  Endoscopic Healing (I) defined as an endoscopic sub-score of ≤ 1.
  The endoscopic sub-score is part of the 3-Component Adapted Mayo score and ranges from 0 - 3, with higher scores indicating more severe disease.
Corticosteroid-free clinical response at Week 12 | Week 12
  Clinical response and achieving a corticosteroid-free status at Week 12 in subjects using oral corticosteroids at the Baseline visit. Clinical response is defined as a decrease from baseline in the 3-Component Adapted Mayo Score of ≥ 2 points and > 30%, with an accompanying decrease in the sub-score for rectal bleeding of ≥ 1 point or an absolute sub-score for rectal bleeding of ≤ 1.
Corticosteroid-free clinical remission at Week 12 | Week 12
  Clinical remission and achieving a corticosteroid-free status at Week 12 in subjects using oral corticosteroids at the Baseline visit. Clinical remission is defined as a stool frequency sub-score of ≤ 1 associated with a decrease ≥ 1 point from baseline, rectal bleeding sub-score of 0, and an endoscopic sub-score of ≤ 1 using the 3-Component Adapted Mayo Score.
Changes from baseline in individual Adapted Mayo sub-scores at Week 12 | Week 12
  The Adapted Mayo Score is a measure of UC disease ranging from 0 to 12 points and consists of 4 sub-scores, each graded from 0 - 3 with higher scores indicating more severe disease. The sub-scores are stool frequency (0 - 3); rectal bleeding (0 - 3); findings of endoscopy (0 - 3); and Physician's Global Assessment [PGA] (0 - 3).

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Responsible Medical Officer, Study Director — Sublimity Therapeutics (HoldCo) Ltd
Locations (89):
- United States (8):
  - Palmtree Clinical Research Inc, Palm Springs, California
  - Advanced Research Institute, Largo, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - Endoscopic Research Inc, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - AGA Clinical Reasearch Associates, LLC, Egg Harbor, New Jersey
  - Baylor College of Medicine, Houston, Texas
  - Biopharma Informatic, LLC., Houston, Texas
- Belarus (3):
  - Grodno Regional Clinical Hospital, Grodno
  - Gomel Regional Clinical Hospital, Homyel
  - City Clinical Emergency Hospital, Minsk
- Bulgaria (3):
  - MedConsult Pleven, Pleven
  - Medical Center Asklepion, Sofia
  - UMBAL Tsaritsa Joanna ISUL, Sofia
- Canada (2):
  - Dalhousie University - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
- France (4):
  - CHU Amiens Picardie - Service Hépato-Gastroentérologie, Amiens
  - CHU DE MONTPELLIER - Hôpital St ELOI, Montpellier
  - CHU de Saint-Etienne - Service de Gastro-Entérologie-Hépatologie, Saint-Etienne
  - Hôpital de Brabois Service d'Hépato-Gastro-Entérologie, Vandœuvre-lès-Nancy
- Germany (9):
  - Eugastro GmbH, Leipzig, Saxony
  - Medizinische Klinik für Gastroenterologie, Infektiologie, Rheumatologie charite, Berlin
  - Krankenhaus Walfriede, Akademisches Lehrkrankenhaus der Charite, Berlin
  - Klinik für Gastroenterologie, Pulmologie und allg. lnnere Medizin, Cologne
  - Agaplesion Markus Krankenhaus Medizinischen Klinik I, Gastroenterologie, Hepatologie, Onkologie, lnfektiologie, Frankfurt
  - Universitatsklinikum Freiburg, Medizinische Klinik, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Zentrym für Innere Medizin, Hanover
  - Universität Leipzig, Klinik f. Gastroenterologie und Rheumatologie, Leipzig
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
- Hungary (4):
  - DRC Gyógyszervizsgáló Központ Kft., Balatonfüred
  - Semmelweis University, Budapest
  - Semmelweis University, AOK Varosmajori Sziv- es Ergyogyaszati Klinika,, Budapest
  - Bugat Pal Hospital, Gyöngyös
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
- Israel (4):
  - Gastroenterology Institute, Emek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Clalit Health Services Jerusalem, Jerusalem
  - Institute of Gastroenterology, Meir Medical Center, Kfar Saba
- Italy (5):
  - Humanitas Research Hospital, IBD Center, Milan
  - A.0.U. di Modena - Policlinico S.C. di Gastroenterologia, Modena
  - Fondazione IRCCS Policlinico San Matteo - Medicina Generale I, Pavia
  - ASST Rhodense - Ospedale di Rho, Rho
  - Fondazione Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Poland (6):
  - Centrum Opieki Zdrowotnej Orkan-med, Ksawerów
  - Oddział Kliniczny Gastroenterologii Ogólnej i Onkologicznej SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego UM, Lodz
  - Medicome Sp. z o.o., Oświęcim
  - Centrum Medyczne Medyk, Rzeszów
  - Endoskopia sp. z o.o., Sopot
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
- Romania (3):
  - MedLife Grivita, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - University Hospital Bucharest, Bucharest
- Russia (10):
  - Federal State Center of Coloproctology, Moscow
  - LLC Medical center Healthy family, Novosibirsk
  - Military Medical Academy, Saint Petersburg
  - North-Western State Medical University n.a. I.I.Mechnikov, Saint Petersburg
  - Saint-Petersburg State Medical Academy n.a. I.I. Mechnikov of Federal Agency of Healthcare & Social Development, Saint Petersburg
  - Scientific Research Center Eco-Safety LLC, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Non state Public Health Institution "Railway clinical hospital on station Samara" of joint stock company Russian railways, Samara
  - Saratov State Medical University, Saratov
  - Siberia State Medical University, Tomsk
- Serbia (4):
  - Clinical Center Zvezdara, Belgrade
  - Clinical Hospital Center "Dr Dragisa Misovic-Dedinje", Belgrade
  - Clinical-Hospital Centre Bezanijska Kosa - Gastroenterology Department, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- Hospital Universitario Virgen de la Macarena, Seville, Spain
- Ukraine (14):
  - Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Ivano-Frankivsk National Medical University, Regional Clinical Hospital, Ivano-Frankivsk
  - Kharkiv City Clinical Hospital No 2 n.a. prof. O.O.Shalimov, Kharkiv
  - Kiev City Clinical Hospital No. 1, Kiev
  - Communal Institution of Kyiv Regional Council "Kyiv Regional Clinical Hospital", Kyiv
  - Ukrainian-German Gastroenterology Center "BYK-Kyiv", Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Communal Nonprofit Enterprise "Lviv Clinical Emergency Care Hospital", Lviv
  - Communal Nonprofit Entreprise, "Lviv Clinical Emergency Care Hospital", 1st Therapeutic Dpt, Lviv
  - Communal Nonprofit Enterprise "Odesa Regional Clinical Hospital", Odesa
  - Communal Nonprofit Enterprise "Ternopil University Hospital" of Ternopil Regional Council, Ternopil
  - Municipal Institution "Uzhhorod Central District Hospital", Uzhhorod
  - Medical Center "Health Clinic", Vinnytsia
  - Communal Non-profit Enterprise "Vinnytsia City Clinical Hospital #1", Vinnytsia
- United Kingdom (7):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - South Eastern Health & Social Care Trust, Ulster Hospital, Belfast, Co Antrim
  - Royal Liverpool & Broadgreen University Hospitals NHS Trust, Liverpool, Merseyside
  - Queen Elizabeth Hospital Birmingham, University Hospitals Birmingham NHS Foundation Trust, Birmingham, Warwickshire
  - Barnsley Hospital NHS Foundation Trust, Barnsley, Yorkshire
  - University College London Hospital NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided